CLINICAL TRIAL: NCT05933083
Title: MCNAIR Study: coMparative effeCtiveness of iN-person and teleheAlth cardIac Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Mayo Clinic (Other); University of Michigan (Other); University of Pittsburgh (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IHS-2021C3-24147
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Myocardial Infarction; Heart Failure, Systolic; Heart Valve Diseases; Angina, Stable; Coronary Artery Disease; Heart Transplant
Keywords: cardiac rehabilitation, telehealth
MeSH Terms: conditions — Myocardial Infarction; Heart Failure, Systolic; Heart Valve Diseases; Angina, Stable; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person cardiac rehabilitation (Active Comparator): Participants will participate in 12-week in-person cardiac rehabilitation as delivered at the site where they are enrolled. The typical course is 36 sessions of group exercise, health education, and counseling over 12 weeks.
  Interventions: Behavioral: In-person cardiac rehabilitation
- Telehealth cardiac rehabilitation (Active Comparator): Participants will participate in 12-week telehealth cardiac rehabilitation. The program will follow the same core components as in-person cardiac rehabilitation, but in-person supervised exercise will not be required. The core element of telehealth cardiac rehabilitation is 12 weekly individual telehealth sessions between the patient and cardiac rehabilitation provider.
  Interventions: Behavioral: Telehealth cardiac rehabilitation

INTERVENTIONS:
Behavioral: In-person cardiac rehabilitation — In-person exercise training, health education, and counseling
  Arms: In-person cardiac rehabilitation
Behavioral: Telehealth cardiac rehabilitation — Telehealth exercise training, health education, and counseling
  Arms: Telehealth cardiac rehabilitation

SUMMARY:
Cardiac rehabilitation is a medically recommended program for patients with certain heart conditions. It includes exercise training, health education, and counseling. Unfortunately, many patients do not participate in cardiac rehabilitation. Some find it challenging to attend the in-person sessions. This study aims to compare two methods of delivering cardiac rehabilitation: in-person and through telehealth. The investigators want to know if the effects of these two programs are alike and if certain individuals benefit more from one program over the other.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Eligible for cardiac rehabilitation

   1. Diagnosis within 1 year prior to consent

      * Myocardial infarction
      * Percutaneous coronary intervention
      * Coronary artery bypass
      * Heart valve repair or replacement
      * Heart transplant
   2. Chronic stable angina, or
   3. Chronic systolic heart failure (ejection fraction ≤ 35%)
   4. Referred to cardiac rehabilitation by a doctor or advanced practice provider for another indication that is covered by the participant's insurance, such as heart failure with preserved ejection fraction or aortic surgery.
3. Willing to be randomized to in-person or telehealth cardiac rehabilitation
4. Able to communicate in English or Spanish

Exclusion Criteria:

1. Unstable arrhythmias which may make unmonitored exercise unsafe (e.g., history of ventricular tachycardia not on medical therapy and without an implantable cardioverter defibrillator)
2. Unsafe for patient to participate in the opinion of the investigator
3. Hospice
4. Unable to consent for self

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Change in six minute walk distance | Baseline and 12 months
  The distance walked in six minute on a standard course will be measured in meters at baseline and 12 months.

SECONDARY OUTCOMES:
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health 10 Scores - Mental Health | Baseline and 12 months
  A change in PROMIS Global Health 10 scores will be measured during the first 12 months of the study. The PROMIS Global Health 10 questionnaire is a self-assessed questionnaire that asks participants to respond to 10 questions with a 5-point ordinal rating scale of "Never," "Rarely," "Sometimes," "Often," and
Change in PROMIS Global Health 10 Scores - Physical Health | Baseline and 12 months
  A change in PROMIS Global Health 10 scores will be measured during the first 12 months of the study. The PROMIS Global Health 10 questionnaire is a self-assessed questionnaire that asks participants to respond to 10 questions. The physical health subscale consists of four questions with a raw score between 4 and 20 that is converted to a standardized T-score. Higher scores represent better physical health.
Change in Generalized Anxiety Disorder (GAD)-7 | Baseline and 12 months
  A change in GAD-7 scores will be measured during the first 12 months of the study. The GAD-7 questionnaire is a self-assessed questionnaire that asks participants to respond to 7 questions with response option scores ranging from 0 to 3. The scale ranges from 0 to 21. Higher scores represent more anxiety symptoms.
Change in Patient Health Questionnaire (PHQ)-9 | Baseline and 12 months
  A change in PHQ-9 scores will be measured during the first 12 months of the study. The PHQ-7 questionnaire is a self-assessed questionnaire that asks participants to respond to 9 questions with response option scores ranging from 0 to 3. The scale ranges from 0 to 27. Higher scores represent more depressive symptoms.
Blood pressure control | 12 months
  Blood pressure less than 130/80 mmHg
Participation in cardiac rehabilitation | 12 months
  Participation in CR, defined as proportion of core sessions attended (out of 36 sessions for in-person and 12 sessions for telehealth)
Survival free of hospitalization for myocardial infarction, heart failure, or stroke/TIA. | 24 months
Change in PROMIS Global Health 10 Scores - Mental Health | Baseline and 3 months
  A change in PROMIS Global Health 10 scores will be measured during the first 3 months of the study. The PROMIS Global Health 10 questionnaire is a self-assessed questionnaire that asks participants to respond to 10 questions . The mental health subscale consists of four questions with a raw score between 4 and 20 that is converted to a standardized T-score. Higher scores represent better mental health.
Change in PROMIS Global Health 10 Scores - Mental Health | Baseline and 24 months
  A change in PROMIS Global Health 10 scores will be measured during the first 24 months of the study. The PROMIS Global Health 10 questionnaire is a self-assessed questionnaire that asks participants to respond to 10 questions . The mental health subscale consists of four questions with a raw score between 4 and 20 that is converted to a standardized T-score. Higher scores represent better mental health.
Change in PROMIS Global Health 10 Scores - Physical Health | Baseline and 3 months
  A change in PROMIS Global Health 10 scores will be measured during the first 3 months of the study. The PROMIS Global Health 10 questionnaire is a self-assessed questionnaire that asks participants to respond to 10 questions. The physical health subscale consists of four questions with a raw score between 4 and 20 that is converted to a standardized T-score. Higher scores represent better physical health.
Change in PROMIS Global Health 10 Scores - Physical Health | Baseline and 24 months
  A change in PROMIS Global Health 10 scores will be measured during the first 24 months of the study. The PROMIS Global Health 10 questionnaire is a self-assessed questionnaire that asks participants to respond to 10 questions. The physical health subscale consists of four questions with a raw score between 4 and 20 that is converted to a standardized T-score. Higher scores represent better physical health.
Change in GAD-7 | Baseline and 3 months
  A change in GAD-7 scores will be measured during the first 3 months of the study. The GAD-7 questionnaire is a self-assessed questionnaire that asks participants to respond to 7 questions with response option scores ranging from 0 to 3. The scale ranges from 0 to 21. Higher scores represent more anxiety symptoms.
Change in GAD-7 | Baseline and 24 months
  A change in GAD-7 scores will be measured during the first 24 months of the study. The GAD-7 questionnaire is a self-assessed questionnaire that asks participants to respond to 7 questions with response option scores ranging from 0 to 3. The scale ranges from 0 to 21. Higher scores represent more anxiety symptoms.
Change in PHQ-9 | 3 months
  A change in PHQ-9 scores will be measured during the first 3 months of the study. The PHQ-7 questionnaire is a self-assessed questionnaire that asks participants to respond to 9 questions with response option scores ranging from 0 to 3. The scale ranges from 0 to 27. Higher scores represent more depressive symptoms.
Change in PHQ-9 | 24 months
  A change in PHQ-9 scores will be measured during the first 24 months of the study. The PHQ-7 questionnaire is a self-assessed questionnaire that asks participants to respond to 9 questions with response option scores ranging from 0 to 3. The scale ranges from 0 to 27. Higher scores represent more depressive symptoms.
Blood pressure control | 3 months
  Blood pressure less than 130/80 mmHg
Blood pressure control | 24 months
  Blood pressure less than 130/80 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Beatty, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (5):
- United States (5):
  - University of California, San Francisco, San Francisco, California
  - Denver Health, Denver, Colorado
  - Johns Hopkins University Medical Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
After study completion, the investigators will generate a de-identified dataset that may be shared with other researchers upon request.